CLINICAL TRIAL: NCT06701578
Title: The Effect of the Safe and Sound Protocol on Depression and Anxiety Symptoms
Acronym: SSP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A24-341
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depression
Keywords: auditory; sound
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe and Sound Protocol Group (Experimental): The intervention involves listening to specially designed filtered and modulated music that is tailored to enhance the individual's auditory system's ability to process and respond to auditory stimuli.
  Interventions: Other: Safe and Sound Protocol
- Control Group (Placebo Comparator): The control condition involves listening to music that is not filtered and modulated.
  Interventions: Other: Control

INTERVENTIONS:
Other: Safe and Sound Protocol — Listening to specially designed filtered and modulated music that is tailored to enhance the individual's auditory system's ability to process and respond to auditory stimuli for up to five hours.
  Arms: Safe and Sound Protocol Group
Other: Control — Listening to music that is not filtered and modulated for up to five hours.
  Arms: Control Group

SUMMARY:
The goal of this study is to determine if a developed protocol involving modulated auditory stimulation is better than non-modulated auditory stimulation in reducing anxiety and depression in human subjects.

DETAILED DESCRIPTION:
A protocol has been developed that provides patients an intervention of listening to specifically designed filtered and modulated music that stimulates the part of the nervous system that induces a calm physiological (bodily) state. This enhancement may help re-establish nerve pathways between auditory processing and emotional regulation systems which promotes improved emotional regulation in regards to depression and anxiety. For this study, participants will either be assigned to the active group who receives the therapy with auditory stimulation that is modulated, or be assigned to the control group who will receive the same interventions without the modulated auditory stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Client of DayBridge
* 18 years old or older
* Meet the DMS-V diagnostic criteria of Major Depressive Disorder and/or Generalized Anxiety Disorder

Exclusion Criteria:

* Previous participation in the SSP
* Self-reported hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | 10 minutes at enrollment visit and 10 minutes at final study visit 3 weeks after enrollment
  The 9-question Patient Health Questionnaire (PHQ-9) is a self-report screening tool for adults in primary care settings for assessing the presence and severity of depression symptoms. Items are aligned with the DSM-5 diagnostic criteria for MDD and queries the individual's experience in the past two weeks. Likert-type responses range from 0 ("Not at all") to 3 ("Nearly every day"). Good reliability and validity have been demonstrated. The PHQ-9 score is the key outcome variable for MDD symptoms.
  The total score is obtained by summing the values of the seven items. The total score ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
GAD-7 | 10 minutes at enrollment visit and 10 minutes at final study visit 3 weeks after enrollment.
  The Generalized Anxiety Disorder 7 (GAD 7) is a self-administered measure of the frequency and severity of generalized anxiety disorder symptoms based on seven DSM-5 diagnostic criteria for GAD. It is typically used in outpatient and primary care settings. Response options are a Likert-type scale ranging from 0 ("Not at all") to 3 ("Nearly every day"). An additional question is a global rating of the severity of the patient's anxiety over the past 2 weeks. The measure is considered sensitive and has shown adequate internal consistency reliability and validity for assessing anxiety across a wide range of samples and settings. The GAD-7 score is the key outcome variable for GAD symptoms.
  The scoring involved summing the values of all seven items to obtain a score between 0 and 21. Higher scores indicate greater severity of anxiety symptoms.
BPQ-SF | 10 minutes at enrollment visit and 10 minutes at final study visit 3 weeks after enrollment.
  The Body Perception Questionnaire - Short Form (BPQ-SF) is an abbreviated version of the original self-report measure of body awareness and autonomic reactivity. The questionnaire consists of two subscales, Body Awareness (26 items) and Autonomic Nervous System Reactivity (20 items). The Likert-type scale answers range from 1 ("Never") to 5 ("Always"). Total scores for each subscale, which are key outcome variables, are summed and compared to T-scores in the BPQ Manual.
Heart Period and Respiratory Sinus Arrhythmia | 10 minutes at enrollment visit and 10 minutes at final study visit 3 weeks after enrollment.
  Heart period will be recorded at 1000 Hz using a Polar H10 chest strap device. This device has shown strong agreement and small bias compared to electrocardiogram (ECG) recordings. It has been chosen as it is minimally invasive and easy for participants to put on.
  RSA and heart period will be used to calculate the vagal contribution to regulation of the heart, i.e., vagal tone.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Leal, Principal Investigator
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with external entities outside of aggregate form for publication. Deidentified data will be shared with the study sponsor. Study identifiers will be destroyed after publication.

REFERENCES:
- [Background] Using the Safe and Sound Protocol (SSP) in clinical practice-Improving outcomes for clients with sensory processing difficulties and trauma-related challenges. International Journal of Environmental Research and Public Health
- [Background] Vargas S, Lucker JR. A Quantitative Summary of The Listening Program (TLP) Efficacy Studies: What Areas Were Found to Improve by TLP Intervention? Occup Ther Int. 2016 Jun;23(2):206-17. doi: 10.1002/oti.1425. Epub 2016 Feb 17. PMID 26890280
- [Background] Strawn JR, Geracioti L, Rajdev N, Clemenza K, Levine A. Pharmacotherapy for generalized anxiety disorder in adult and pediatric patients: an evidence-based treatment review. Expert Opin Pharmacother. 2018 Jul;19(10):1057-1070. doi: 10.1080/14656566.2018.1491966. PMID 30056792
- [Background] Social Outcomes of a Child with Autism Spectrum Disorder Following a Listening Protocol. Journal of Occupational Therapy, Schools, & Early Intervention
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] A Pilot Study of Integrated Listening Systems for Children With Sensory Processing Problems. Journal of Occupational Therapy, Schools, & Early Intervention
- [Background] Schaffarczyk M, Rogers B, Reer R, Gronwald T. Validity of the Polar H10 Sensor for Heart Rate Variability Analysis during Resting State and Incremental Exercise in Recreational Men and Women. Sensors (Basel). 2022 Aug 30;22(17):6536. doi: 10.3390/s22176536. PMID 36081005
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Meuret AE, Tunnell N, Roque A. Anxiety Disorders and Medical Comorbidity: Treatment Implications. Adv Exp Med Biol. 2020;1191:237-261. doi: 10.1007/978-981-32-9705-0_15. PMID 32002933
- [Background] Mahlich J, Tsukazawa S, Wiegand F. Estimating Prevalence and Healthcare Utilization for Treatment-Resistant Depression in Japan: A Retrospective Claims Database Study. Drugs Real World Outcomes. 2018 Mar;5(1):35-43. doi: 10.1007/s40801-017-0126-5. PMID 29185233
- [Background] Clinical effectiveness of the Safe and Sound Protocol in improving sensory processing: A pilot study. Frontiers in Psychiatry
- [Background] Kawai H, Kishimoto M, Okahisa Y, Sakamoto S, Terada S, Takaki M. Initial Outcomes of the Safe and Sound Protocol on Patients with Adult Autism Spectrum Disorder: Exploratory Pilot Study. Int J Environ Res Public Health. 2023 Mar 9;20(6):4862. doi: 10.3390/ijerph20064862. PMID 36981773
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Domschke K, Stevens S, Pfleiderer B, Gerlach AL. Interoceptive sensitivity in anxiety and anxiety disorders: an overview and integration of neurobiological findings. Clin Psychol Rev. 2010 Feb;30(1):1-11. doi: 10.1016/j.cpr.2009.08.008. PMID 19751958